CLINICAL TRIAL: NCT05736120
Title: Persons With Obesity (PwO) Exploratory Research - India
Brief Title: Persons With Obesity (PwO) Exploratory Research
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-7679; U1111-1285-1486 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase I: Online bulletin boards (OBB)
  Interventions: Other: No treatment given
- Phase II: Virtual focus groups (real-time)
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
The purpose of this study is to understand the personal flow along the weight loss management journey. A range of variables will be addressed in a survey to explore the weight loss journey, barriers and management. Topics include weight loss strategies and challenges, HCP involvement, and perceptions towards weight loss medications.

Potential participants will be recruited using various online panels. Study participants will be recruited to participate in 2 types of qualitative research.

Phase I: Online bulletin boards (OBB) Phase II: Virtual focus groups (real-time)

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, age above or equal to 18 years at the time of signing informed consent.
3. Current body mass index (BMI) of 25 or greater
4. Not currently pregnant
5. Does not participate in intense fitness or body building program
6. Weight loss not through illness or injury
7. At least somewhat concerned about current weight
8. If no plans for weight loss in the next six months, has made at least 1 weight loss effort in last 5 years
9. Struggling with weight for at least 3 years

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study
2. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
3. Does not meet inclusion criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited to participate in 2 types of qualitative research. Online Bulletin Boards and Virtual Focus Groups
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-02-19 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Description of perceptions, behaviours and awareness related to obesity and obesity management among people living with obesity. | 5 days (Phase 1)
  120-minute OBB discussion with numeric and open-ended response (Phase 1)
Description of perceptions, behaviours and awareness related to obesity and obesity management among people living with obesity. | 1 day (Phase 2)
  90-minute focus group with open-ended response (Phase 2)
Assessment of triggers for people with obesity to request medical therapy and expectations for both therapy available and their weight loss journey. | 5 days (Phase 1)
  120-minute OBB discussion with numeric and open-ended response (Phase 1)
Assessment of triggers for people with obesity to request medical therapy and expectations for both therapy available and their weight loss journey. | 1 day (Phase 2)
  90-minute focus group with open-ended response (Phase 2)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bengaluru, India

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com